CLINICAL TRIAL: NCT01356212
Title: Scintigraphic Assessment of Nasal Deposition and Clearance of 99mTc DTPA Ketorolac Solution Administered Using the Valois Nasal Spray Device
Brief Title: Assessment of Nasal Deposition and Clearance of Ketorolac Solution Administered Using the Valois Nasal Spray Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROX 2002-02
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Ketorolac Tromethamine

ARMS (3):
- Regimen A: Ketorolac tromethamine (Gentle Sniff - Upright) (Experimental): Gentle sniff-inhalation with the volunteer upright for dosing and imaging
  Interventions: Drug: Ketorolac tromethamine
- Regimen B: Ketorolac tromethamine (Vigorous Sniff - Upright) (Experimental): Vigorous sniff-inhalation with the volunteer upright for dosing and imaging
  Interventions: Drug: Ketorolac tromethamine
- Regimen C: Ketorolac tromethamine (Gentle Sniff - Semi-supine) (Experimental): Gentle sniff-inhalation with the volunteer semi-supine for dosing and imaging
  Interventions: Drug: Ketorolac tromethamine

INTERVENTIONS:
Drug: Ketorolac tromethamine — 30 mg ketorolac (15 mg (100 ul) per nostril) administered intranasally
  Arms: Regimen A: Ketorolac tromethamine (Gentle Sniff - Upright)
Drug: Ketorolac tromethamine — 30 mg ketorolac (15 mg (100 ul) per nostril) administered intranasally
  Arms: Regimen B: Ketorolac tromethamine (Vigorous Sniff - Upright)
Drug: Ketorolac tromethamine — 30 mg ketorolac (15 mg (100 ul) per nostril) administered intranasally
  Arms: Regimen C: Ketorolac tromethamine (Gentle Sniff - Semi-supine)

SUMMARY:
This was a randomised three-way crossover design study. The study consisted of three study periods each separated by a minimum 44 hour washout period. During the course of each study period, scintigraphic images were acquired at planned intervals after dosing. Subjects were able to leave the clinical unit after the completion of study specific procedures at 6 hours post-dose.

The primary objective of the study was to determine whether any of the radiolabelled ketorolac formulation was deposited in the lungs of healthy volunteers following nasal inhalation under three different conditions (gentle sniff-inhalation with subject standing, vigorous sniff-inhalation with subject standing, gentle sniff-inhalation with subject semi-supine). The secondary objectives were to determine the deposition pattern of radiolabelled ketorolac solution in the nasal cavity, and clearance of the radiolabel over a six-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating, surgically sterile or post-menopausal females (post-menopausal was defined as > 2 years post-last period and more than 50 years of age), or using an acceptable form of contraception as defined in section 9.3.2 (g)
* Aged 18-65 years
* Body Mass Index of between 18 and 30 kg/m2

Exclusion Criteria:

* Participation in a clinical research study involving investigational drugs or dosage forms within the previous 4 months
* Subjects who had sought advice from their GP or consulted a counsellor for abuse or misuse of alcohol, non-medical, medicinal drugs, or other substance-abuse such as solvents. Any current or past use of Class A drugs such as opiates, ecstasy, LSD, and amphetamines (Class B). Volunteers that admitted to past use of cannabis were not excluded as long as they had a negative drugs of abuse test and had been abstinent for at least 12 months
* Positive drugs of abuse test result
* Regular alcohol consumption in males >21 units per week and females >14 units per week. (one unit of alcohol was defined as 0.5 pint (280 ml) of beer or cider, 1 glass (125 ml) wine, 1 glass (70 ml) of sherry or port, 1 measure (25 ml) of whisky, brandy or rum. For low alcohol drinks, one unit of alcohol was defined as 2 glasses (250 ml) of low alcohol wine and 5 half pints (840 ml) of low alcohol beer)
* Current smokers, i.e. those who had smoked within the last 12 months
* A breath carbon monoxide reading of greater than 10 ppm either at the pre-study medical examination or on a study day prior to dosing
* Females of child bearing potential who were sexually active and either not surgically sterile, post-menopausal or not using a form of acceptable contraceptive (contraceptive pills/injection, condoms with spermicide, IUCDs (coils) and diaphragms with spermicide (only if the woman was 35 or more) or abstinence
* Radiation exposure from clinical trials, including that from the present study and from diagnostic X-rays but excluding background radiation, exceeding 5 mSv in the last twelve months or 10 mSv in the last five years. No subject whose occupational exposure is monitored will participate in the study
* Clinically significant abnormal biochemistry, haematology or urinalysis
* Screening FEV1 < 80% of the predicted value for their age, sex, height and race
* History of chronic respiratory disorders or bronchospasm
* History of adverse reaction or allergy to ketorolac or di-sodium EDTA
* History of severe or multiple allergies, including hayfever and perennial rhinitis
* History of adverse reaction or allergy to aspirin or any other non-steroidal anti inflammatory drug (e.g., ibuprofen, flurbiprofen, ketoprofen or diclofenac)
* History of infantile bronchiolitis, or a history or the presence of asthma, or wheezy respiration, hayfever and perennial rhinitis
* History of nasal fracture, nasal deformity or nasal polyps
* History of disease, surgery, or abnormality of the upper respiratory tract, especially the nasal cavity
* History of significant nose bleeds
* Sinusitis within four weeks of the first study period
* Nasal jewelry or nasal piercings
* Subjects using topical nasal medication e.g. decongestants, within 14 days prior to the first dosing day
* Upper respiratory tract infection (excluding otitis media) within 14 days of the first study day, or lower respiratory tract infection within the previous 3 months
* Subjects taking any medication that might affect the respiratory tract within 14 days of the first study day
* Non-prescription and prescription medication (including vitamins and natural or herbal remedies eg. St Johns Wort) within 14 days of the first study day (oral contraceptives, contraceptive implants or depot injections, intra-uterine devices with hormonal implants, Hormone Replacement Therapy (HRT) and occasional paracetamol (up to 4 g daily) were permitted)
* History of peptic ulceration or gastrointestinal bleeding
* History of kidney disease
* History of clotting disorders
* Failure to satisfy the Principal Medical Investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-09; Primary Completion 2002-10 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Scintigraphic images of radiolabeled ketorolac solution entering the lungs and subsequently being cleared from the lungs following administration to the nostrils using a Valois nasal device. | Change from baseline to immediately post-dose, 10, 20, 30, 45, and 60 minutes and 2, 4, and 6 hours post dose

SECONDARY OUTCOMES:
Scintigraphic assessment of the deposition pattern of radiolabeled ketorolac solution in the nasal cavity, nasopharynx, esophagus, and stomach. | Change from baseline to immediately post-dose, 10, 20, 30, 45, and 60 minutes and 2, 4, and 6 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: L Rankin, MD, Principal Investigator — Pharmaceutical Profiles, Ltd
Locations (1):
- Pharmaceutical Profiles, Ltd, Ruddington, Nottingham, United Kingdom